CLINICAL TRIAL: NCT03152201
Title: I Potenziali Somato-sensoriali Nella Chirurgia Degli Aneurismi Cerebrali
Brief Title: New Findings About Somatosensory Evoked Potentials (SEP) During Surgery for Cerebral Aneurysms
Status: Completed | Type: Observational
Sponsor: Luca Valci (Other)
Responsible Party: Sponsor-Investigator, Luca Valci, Dr. med., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: NCH-2017-01
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electrophysiological signal — trasmit the electrophysiological signals to the neurosurgeon through the hardware

SUMMARY:
During surgery, electrophysiological signals will be acquired with the instrument (ISIS IOM, NeuroExplore, Software Version 4.4, Inomed) already in use at the Neurosurgery Service of the Neurocentro of the Hospital Civic Italian Switzerland in Lugano. Simultaneously to Somatosensorial Evoked Potential (SEP) will also be recorded the Electroencephalography (EEG) activity with the same detection of locations.

For the purposes of the study the signals transmitted to the neurosurgeon through the hardware and the corresponding assessments done by the neurophysiologist responsible for intraoperative monitoring will be recorded. It will also be kept track of procedures performed during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient bearer of a not broken cerebral aneurysm, which has been defined per size and morphology susceptible to surgery
* Aneurysms located on cerebral arteries of the anterior circulation (carotid, middle cerebral arteries, anterior cerebral, anterior communicating, pericallose); Cases of multiple aneurysms are also eligible
* Informed consent for participation in the study

Exclusion Criteria:

* Patient with an aneurysm of the posterior circulation (vertebrobasilar system)
* The aneurysm was a source of bleeding (subarachnoid hemorrhage, intracerebral, intraventricular).
* Patient with a pace-maker (for the risk that the electric currents used in the study could compromise the operation of the pace-maker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient bearer of a not broken cerebral aneurysm
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
hardware performance | at the moment of the surgery
  Collection of information on the hardware performance for reading and interpretation of the SEP and EEG signal and sending an alarm in visual form (light signal) in the eyepiece of the operating microscope during cerebral aneurysm interventions
Identification of sensitive electrophysiological index sensible to cerebral ischemic suffering | up to 3 months
  study of the morphology and the analysis of the high frequency of the SEP signal

CONTACTS AND LOCATIONS:
Overall Officials: Luca Valci, MD, Study Chair — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Neurocentro della Svizzera Italiana (NSI), Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No